CLINICAL TRIAL: NCT05331963
Title: The Effects of Functional Kinesio Taping on Subacromial Space in Athletes With Rotator Cuff Tendinopathy
Brief Title: Effects of Functional Kinesio Taping on Subacromial Space in Athletes With Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01022 Hajra Qureshi
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping with rehabilitation program group (Experimental): Rehabilitation program will be given to this group in addition to Kinesio taping on skin for 72 hour.
  Interventions: Other: Kinesio Taping
- Rehabilitation plan group (No Intervention): The rehabilitation program will be provided individually to all participants (twice weekly during the first 4 weeks, then once weekly)

INTERVENTIONS:
Other: Kinesio Taping — Kinesio tape is designed in a specific way that it mimics the human skin nature. It more or less has the same width as the epidermis layer and can be stretched upto 40% of its resting length.Clinically, kinesio tape (KT) is used both alone and with other physiotherapeutic interventions, mainly for the pain control, to reduce inflammation, and to improve functional activity in patients with shoulder pain
  Arms: Kinesio taping with rehabilitation program group

SUMMARY:
To determine the effects of functional kinesio taping on subacromial space in athletes with rotator cuff tendinopathy.

DETAILED DESCRIPTION:
Subacromial impingement is a condition among athletes those involved in overhead sports activities such as swimming and volleyball. According to Neer there are two main categories of shoulder impingement, these are structural and functional. Structural: caused by reduction of the subacromial space (SAS) due to bony growth, calcification or soft tissue inflammation whereas functional is caused by or superior migration of the humeral head due to muscular weakness imbalance. In some cases subacromial impingement can be result from a combination of both structural and functional factors.Maintenance of the SAS during arm elevation is thus essential for the prevention of Rotator cuff tendinopathy.

The aim of this randomized controlled trial (RCT) is to evaluate the long-term effects of scapular KT, added to a 6-week rehabilitation program, on the subacromial space at different arm positions in athletes with Rotator cuff tendinopathy. To better understand the underlying mechanisms of KT, our secondary objective addressed the effects of KT on reliving pain-free and full ROM of shoulder joint.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 35 years
* Both gender
* Athletes participating in volley ball, tennis, badminton and golf.
* Presence of shoulder pain in abduction and external rotation during training for more than three months
* Three out of five positive results for the following: painful arc, pain or weakness with resisted external rotation, abduction, Neer test, Hawkins Kennedy test, empty can test/Jobe test

Exclusion Criteria:

* H/O shoulder fractures,
* Instability or dislocation (positive apprehension and relocation tests)
* Frozen shoulder (All stages)
* Recent shoulder surgery for a shoulder injury

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Subacrimial space measurement by Ultrasonography | Six weeks
  In order to visualize and measure the subacromial space, the Diagnostic Ultrasound will be used with Aquasonic ultrasound gel as the coupling medium. An ultrasound scanner (Canon aplio i600) with frequency of 1 to 22 MHz curved probe will be used in this study to get images. The probe of US will be placed on the anterior-lateral surface of the acromion process, next to the longitudinal axis of the humeral head, and this is the point likely to view the acromion process and humeral head at the same time. The AHD will then measured from inferior surface of acromion process to the superior surface of the humeral head.The distance is basically from cortical layers of both acromion and humerus bone. The acromio humeral distance will be measured at resting position (0° elevation) of shoulder in millimeters.
Visual Analogue Scale | Six weeks
  This scale consist of 0 to 10 rating in which 0 indicates no pain, and 10 indicates the worst pain.(9) The score of VAS is determined by measuring the distance between the no pain or 0 anchor and to the point where patient draw a mark. A higher score indicates greater pain intensity.
The Disabilities of Arm, Shoulder and Hand Questionnaire | Six weeks
  The DASH will be used to measure functional disorder, physical disability and symptoms of the upper limbs. It consists of 30 questions. 21 questions are related to specific physical tasks in which a person felt difficulty performing last week. 6 questions are to assess specific symptoms including pain, numbness and stiffness. 3 questions are about social and occupational limitations. A 100 point score signifies the most severe disability.
The Western Ontario Rotator Cuff Index | Six weeks
  This instrument consists of 21 items with 5 further categories: i) 6 items of Physical symptoms,ii) 4 items of sports and recreation functions, iii) 4 items of work functions, iv) 4items of lifestyle functions and v) emotional function with 3 items. The instrument has clear instructions to the patients in addition to the explanation of each item of every category.

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, Ph.D., Principal Investigator — Riphah International University
Locations (1):
- Pain and Spine Clinic, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No